CLINICAL TRIAL: NCT07023835
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Usnoflast Administered to Adult Subjects With ALS
Brief Title: Usnoflast Neuromuscular Investigation for Treatment Efficacy in Amyotrophic Lateral Sclerosis
Acronym: UNITE-ALS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USNO.24.002
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis,; ALS; Usnoflast
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 50 mg Usnoflast (Active Comparator): 50 mg Usnoflast capsules and matching placebo of 25 mg capsule under fasting conditions twice a day orally for 36 weeks
  Interventions: Drug: 50 mg Usnoflast
- 75 mg Usnoflast (Active Comparator): 25 mg + 50 mg Usnoflast capsules under fasting conditions twice a day orally for 36 weeks
  Interventions: Drug: 75 mg Usnoflast
- Placebo (Placebo Comparator): Matching placebo of 25 mg and 50 mg under fasting conditions twice a day orally for 36 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg Usnoflast — 50 mg Usnoflast (50 mg Usnoflast capsules and matching placebo of 25 mg capsule)
  Other Names: Not any
  Arms: 50 mg Usnoflast
Drug: 75 mg Usnoflast — 75 mg Usnoflast (25 mg + 50 mg Usnoflast capsules)
  Other Names: Not any
  Arms: 75 mg Usnoflast
Drug: Placebo — Matching placebo of 25 mg and 50 mg
  Other Names: Not any
  Arms: Placebo

SUMMARY:
Usnoflast Neuromuscular Investigation for Treatment Efficacy in Amyotrophic Lateral Sclerosis

DETAILED DESCRIPTION:
A phase 2b, randomized, double-blind, placebo-controlled, parallel-group, multicenter 36 weeks study to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of Usnoflast administered to adult subjects with Amyotrophic Lateral Sclerosis followed by 16 weeks open label extension study.

This Open Label Extension will be a multicenter, 16-week, single arm study to confirm the long-term safety and efficacy of Usnoflast in subjects with ALS. Eligible subjects of all three arms of the main study will be recruited in the OLE phase and will receive Usnoflast (75 mg) for a total of 16 weeks BID (oral capsule administration).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite Amyotrophic lateral sclerosis, according to the revised version of the El Escorial World Federation of Neurology criteria
* Time since onset of first symptom of Amyotrophic lateral sclerosis ≤24 months. Date of Amyotrophic lateral sclerosis symptom onset. For the purposes of this study, the date of symptom onset will be defined as the date the subject first had symptoms of their disease, i.e., limb weakness, dysarthria, dysphagia, shortness of breath, or fasciculations, from the screening visit.
* Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised score of ≥35 at screening.
* Slow vital capacity: ≥60% of predicted capacity at the screening visit.
* Be able to swallow capsules.
* Either not currently receiving riluzole/sodium phenylbutyrate and taurursodiol/tofersen or on a stable dose of riluzole/sodium phenylbutyrate and taurursodiol/tofersen for at least 4 weeks before the screening visit. Subjects receiving riluzole/sodium phenylbutyrate and taurursodiol/tofersen are expected to remain on the same dose throughout the duration of the study.
* Either not currently receiving edaravone or on edaravone treatment. Subjects receiving edaravone must have completed at least 1 cycle of treatment before the screening visit and are expected to continue with a stable dose of edaravone treatment throughout the duration of the study.
* Capable of providing informed consent and complying with study procedures in the opinion of the investigator

Exclusion Criteria:

* Presence of unstable psychiatric disease, cognitive impairment, dementia, or substance abuse that would impair the ability of the subject to provide informed consent, in the opinion of the investigator.
* Serious illness (e.g., pneumonia, septicemia) within 4 weeks of the screening visit; infection requiring hospitalization or treatment with intravenous antibiotics, antivirals, or antifungals within 4 weeks of screening; chronic bacterial infection (such as tuberculosis) deemed unacceptable as per the judgment of the investigator.
* Active herpes zoster infection within 2 months prior to the screening visit.
* Any medical condition that promotes suicidal attempt or behavior within 6 months prior to the screening visit and in the opinion of the investigator might interfere with subject's participation in the study or is a risk for a suicide attempt.
* History of unstable or severe cardiac, pulmonary, oncological, hepatic, or renal disease or active cancer or another medically significant illness other than Amyotrophic lateral sclerosis, precluding safe participation of subject in this study in the opinion of the investigator.
* Known allergy, sensitivity, or intolerance to Investigational product or excipients.
* Subjects who have taken concomitant medications that are substrates of drug metaboliz-ing enzymes (Cytochrome P450 1A2 and/or Cytochrome P450 2B6) within 7 days or 5 half-lives of the medication (whichever is longer) before the first dose of Investigational product and throughout the study.
* Use of any steroids, colchicine, or anti-IL-1 inhibitors within 7 days or 5 half-lives of the medication (whichever is longer) prior to the first dose of Investigational product administration.
* Use of any investigational drug concurrently or within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of Investigational product administration.
* Any clinically significant condition and/or laboratory significant value that would prevent the subject from participating in the study in the opinion of the investigator.
* Received a live vaccine within 14 days before the screening visit or planning to receive during the study duration.
* Subjects who have received stem cell or gene therapy for Amyotrophic lateral sclerosis at any time in the past.
* Following laboratory test values at screening:

  1. Alanine aminotransferase or Aspartate aminotransferase values >3.0 × Upper Limit of Normal
  2. Bilirubin >1.5 × Upper Limit of Normal unless the subject has documented Gilbert's syndrome (isolated bilirubin >1.5 × Upper Limit of Normal is acceptable if bilirubin is fractionated, and direct bilirubin is <35%)
  3. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2
* For those participating in the optional Cerebrospinal fluid collection, contraindications to lumbar puncture including but not limited to lumbar scoliosis, coagulopathy, infection at site of puncture, or use of anticoagulants.
* Subjects with history of epilepsy within 6 months of screening visit.
* Surgery within last 3 months or planned major surgery within next 3 months from the date of screening (other than minor cosmetic surgery and minor dental surgery).
* Use or intended use of any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 4 weeks of screening and up to end of study. Use of such medication will be considered on a case-by-case basis as per the opinion of the investigator and/or independent medical monitor.
* Receiving an elemental diet or parenteral nutrition.
* Received blood transfusion within 3 months prior to screening.
* Subjects with Human immunodeficiency virus, hepatitis B, hepatitis C, coronary artery disease, or active gastrointestinal condition that might interfere with drug absorption.
* Inability to be venipunctured or those not able to tolerate venous puncture.
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of employees of investigator or the investigator.
* Any condition not mentioned in any of above criteria that, as per the investigator, would hinder participation of the subject in the study. This may include, but not limited to, considerations of safety, compliance, or other factors that could impact the integrity of the study or the well-being of the subject.
* If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or of child-bearing potential and unwilling to use effective contraception during the study and for at least 1 month after administration of last dose of Investigational product. If male of reproductive capacity, unwilling to use effective contraception during the study and for at least 1 month after administration of last dose of Investigational product.

For Open Label Extension

Inclusion Criteria:

* Completion in the randomized, double blind Usnoflast study (main study).
* Subjects who elect to continue treatment after completion of Usnoflast phase 2b study must enrol in the OLE within 28 days of the completion of Week 36 visit of the main study.
* Provide a new informed consent to enter the OLE phase.

Exclusion Criteria:

* Discontinued IP prematurely in the double-blind phase of the study for reasons other than tracheostomy or permanent-assisted ventilation.
* Treatment with or use of any restricted medications.
* Any ongoing AE that, in the opinion of the site investigator, is clear contraindication to the IP.
* Unstable cardiac or other life-threatening disease emergent during the randomized, double-blind study
* Any major medical history or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for the study.
* If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or of child-bearing potential and unwilling to use effective contraception during the study and for at least 1 month after administration of last dose of IP. If male of reproductive capacity, unwilling to use effective contraception during the study and for at least 1 month after administration of last dose of IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Usnoflast versus placebo assessed using the revised ALSFRS-R total score | From baseline through Week 36
  Change in disease progression from baseline through Week 36 as measured by ALSFRS-R total score
Efficacy of Usnoflast versus placebo assessed using the survival | From baseline through Week 36
  Change in disease progression from baseline through Week 36 as measured by survival
  Survival is defined based on the time of death or permanent-assisted ventilation (PAV). PAV is defined as the use of invasive or noninvasive mechanical ventilation for >22 hours daily for >7 consecutive days
Effect of Usnoflast versus placebo on survival in Open label extension phase | From baseline through Week 16
  Time from baseline to the occurrence of death or Permanent-assisted ventilation (>22 hours daily for >7 days)
Number of participants with treatment emergent adverse events in open label extension | From baseline through Week 16
  Time from baseline
Number of participants with Serious adverse events in open label extension | From baseline through Week 16
  Time from baseline

SECONDARY OUTCOMES:
Effect of Usnoflast versus placebo on survival | From baseline through Week 36
  Time from baseline to the occurrence of death or Permanent-assisted ventilation (>22 hours daily for >7 days)
Evaluate the effect of Usnoflast versus placebo on Slow vital capacity | from baseline to Week 36
  Change in Slow vital capacity from baseline to Week 36
Evaluate the effect of Usnoflast versus placebo on serum levels of Neurofilament light chain protein | From baseline to Week 36
  Change in serum levels of Neurofilament light chain protein from baseline to Week 36
Evaluate the effect of Usnoflast versus placebo on Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised total score and various functional items/domains of the ALSFRS-R total score | From baseline to Week 36
  To determine the rate of disease progression using the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised total score and scores of various functional items/domains of the ALSFRS-R total score from baseline to Week 36
Evaluate and compare the effect of Usnoflast versus placebo on overall health-related quality of life | From baseline to Week 36
  Change in Amyotrophic Lateral Sclerosis assessment questionnaire-40 (ALSAQ-40) score from baseline to Week 36
Number of participants with treatment emergent adverse events | From baseline to Week 36
  Time from baseline
Number of participants with Serious adverse events | From baseline to Week 36
  Time from baseline
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Peak steady state plasma concentration (Cmax,ss)
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Time to reach peak plasma concentration at steady state (Tmax,ss)
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Accumulation index calculated as a ratio of AUCtau (last dose)/AUCtau (first dose)
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Area under Plasma concentration vs. time curve till the last time point: AUC0-t
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Area under Plasma concentration vs. time curve extrapolated to the infinity: AUC0-∞
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Area under Plasma concentration vs. time curve based on extrapolation: AUCextap
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Elimination rate constant (Kel)
Evaluate Pharmacokinetic of Usnoflast in plasma | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  Elimination half-life (t1/2)
Evaluate Pharmacokinetic of Usnoflast in Cerebrospinal fluid | PK time pts: pre-dose, 2, 4, 6, 8 hours ±30 mins post morning dose at Day 1, Week 16, and Week 36
  The concentration of Usnoflast in CSF.
Effect of Usnoflast versus placebo on Cerebrospinal fluid levels of Neurofilament light chain protein | From baseline to Week 36
  Change in Cerebrospinal fluid levels of Neurofilament light chain protein
To determine the rate of disease progression in open label extension | From baseline to Week 16
  Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised total score and scores of various functional items/domains of the ALSFRS-R total score from baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, Study Director — Zydus Therapeutics Inc.
Locations (17):
- United States (15):
  - Zydus US015, La Jolla, California
  - Zydus US008, Orange, California
  - Zydus US013, San Francisco, California
  - Zydus US005, New Britain, Connecticut
  - Zydus US012, Tampa, Florida
  - Zydus US007, Atlanta, Georgia
  - Zydus US010, Boston, Massachusetts
  - Zydus US006, Detroit, Michigan
  - Zydus US014, Lincoln, Nebraska
  - Zydus US003, Winston-Salem, North Carolina
  - Zydus 009, Pittsburgh, Pennsylvania
  - Zydus US001, Dallas, Texas
  - Zydus US002, Houston, Texas
  - Zydus US004, Richmond, Virginia
  - Zydus US011, Seattle, Washington
- Canada (2):
  - Zydus 101, Toronto, Ontario
  - Zydus 100, Québec, Quebec